CLINICAL TRIAL: NCT06393075
Title: Effect of Preoperative Combined Care Guidance on Pain, Anxiety and Joint Range of Motion in Patients Undergoing Total Knee Arthroplasty
Brief Title: The Effectiveness of Combined Care for Knee Replacement Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-08-016AC
Record Dates: First submitted 2024-04-19; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Arthroplasty, Knee Replacement
Keywords: Total knee replacement; pain scores; anxiety levels; joint mobility

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined care guidance (Experimental): Pain care guidance animation Rehabilitation exercise guidance animation Demonstrate how to perform rehabilitation exercises Demonstrate how to use a walker
  Interventions: Behavioral: combined care guidance
- general care guidance (Active Comparator): Verbal explanation of pain and rehabilitation exercise instructions after surgery
  Interventions: Behavioral: general care guidance

INTERVENTIONS:
Behavioral: combined care guidance — Pain care guidance animation Rehabilitation exercise guidance animation Demonstrate how to perform rehabilitation exercises Demonstrate how to use a walker
  Arms: combined care guidance
Behavioral: general care guidance — general care guidance
  Arms: general care guidance

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of combined care guidance and general care guidance on pain scores, anxiety levels and joint mobility in patients undergoing total artificial knee replacement. The main questions it aims to answer are:

* Does combined care coaching reduce patient pain scores and anxiety levels after surgery?
* Does combined care guidance improve knee joint mobility after surgery? Researchers will compare combined care guidance and general care to see if combined care guidance reduces patients' pain scores and anxiety levels after surgery, and improves knee joint mobility after surgery.

Participants will:

* Watch pain and rehabilitation exercise guidance videos before surgery and learn how to use a walker.
* Complete questionnaires before surgery, 24 hours, 48 hours, 72 hours and three months after surgery.
* Questionnaire records pain level, anxiety level and joint mobility.

DETAILED DESCRIPTION:
Background:The population is aging rapidly, and an aging society is approaching. According to Taiwan government statistics, the population over 65 years old has reached 16.2%. The number of people suffering from knee osteoarthritis has reached 860,000, and the number of patients undergoing total artificial knee replacement has reached 29,000. people.Artificial knee replacement can effectively relieve joint pain, correct joint deformities, and improve joint function. However, patients who undergo total artificial knee replacement still experience moderate to severe pain after surgery. Effective pain control can promote early rehabilitation and early ambulation of patients. In clinical practice, it is more common to provide a single interventional measure to improve the pain level after surgery, but less to provide combined measures before surgery, which leads to the motivation for discussion.

Purpose:To compare the effectiveness of combined care guidance and general care Method:guidance on pain scores, anxiety levels and joint mobility of patients undergoing total artificial knee replacement before surgery, 24 hours, 48 hours, 72 hours and three months after surgery.Experimental group: Researchers provided combined care, watched animated videos, demonstrated rehabilitation exercises and practiced walking using walkers.Control group: The researchers provided general preoperative care and demonstrated rehabilitation exercises and the use of walking aids after surgery.

:This study adopted an experimental research design, single-blind, and randomly assigned groups, one experimental group and one control group.Data were collected five times in total, before surgery, 24 hours after surgery, 48 hours after surgery, 72 hours after surgery and 3 months after surgery.All five data collections are required to fill in the Numerical Rating Scale (NRS) state-trait anxiety inventory (STAI), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)

ELIGIBILITY:
Inclusion Criteria:

* Those who are 20 years old or above (inclusive), have undergone unilateral total knee replacement for the first time, have clear consciousness, can speak Mandarin and Taiwanese, have elementary school-level reading ability, and are willing to participate in the study

Exclusion Criteria:

* Patients with bilateral total knee replacement, osteoarthritis tumors, rheumatoid arthritis, who are unable to cooperate with interventional measures, patients with dementia or cognitive dysfunction who are unable to cooperate; those who are participating in other pain control studies

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
pain scores | baseline, 24 hours, 48 hours, 72 hours and three months after surgery
  Using the Numerical Rating Scale to assess postoperative pain in patients undergoing knee replacement surgery.0 points are not painful, 10 points are the most painful.
anxiety levels | baseline, 24 hours, 48 hours, 72 hours and three months after surgery
  Assessing Anxiety Levels After Knee Replacement Using the State-Trait Anxiety Inventory.Scale scores range from 20 to 80, with lower scores indicating less severe anxiety, 20-39 indicating mild anxiety, 40-59 indicating moderate anxiety, and 60-80 indicating severe anxiety.
joint mobility | baseline, 24 hours, 48 hours, 72 hours and three months after surgery
  Assessment of range of motion after knee surgery using the Western Ontario and McMaster Universities Osteoarthritis Index.

CONTACTS AND LOCATIONS:
Overall Officials: LI YING-HUNG, 32, Principal Investigator — Employment relationship
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan